CLINICAL TRIAL: NCT02386319
Title: Anxiolytic and Analgesic Effects of Melatonin: A Randomized, Double-blinded, Placebo-controlled Clinical Study
Brief Title: Anxiolytic and Analgesic Effects of Melatonin
Acronym: ANAN-Melatonin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Dennis Bregner Zetner, MD Ph d fellow, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Melatonin1234
Record Dates: First submitted 2015-02-24; First posted 2015-03-11 (Estimated); Results first posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Anxiety
Keywords: Melatonin; Surgery; Pharmacokinetic; Anxiolytic
MeSH Terms: conditions — Anxiety Disorders | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin (Active Comparator): Melatonin 10 mg, gelatin capsules. Pharmacokinetic study: 10 mg x 2. In the morning before surgery and in the evening after surgery.
  Anxiolytic and analgesic study: 10 mg x 4. Evening the day before surgery, the morning before surgery, immediately after surgery and the evening after surgery.
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): Gelatin capsules. Anxiolytic and analgesic study. Evening the day before surgery, the morning before surgery, immediately after surgery and the evening after surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — Gelatin capsules
  Arms: Melatonin
Drug: Placebo — Placebo capsules
  Arms: Placebo

SUMMARY:
The study's main objective is to investigate melatonin's anxiolytic and sleep-regulating effects in patients undergoing surgery. Moreover, the investigators intend to investigate the pharmacokinetic parameters of melatonin in this patient population.

DETAILED DESCRIPTION:
The study is separated into two parts. In the first part the patients are undergoing cosmetic breast surgery, and in the second part the patient undergo inguinal og umbilical surgery.

The first part is a cohort at 12 patients undergoing breast surgery. All patients in this group will be treated with melatonin, and the investigators intend to investigate the pharmacokinetic parameters of melatonin. Melatonin will be administrated 60 min. before surgery and the evening after surgery at 9 pm.

All patients will receive an intravenous catheter. The intravenous catheter will be used for blood sampling. A baseline blood sample will be taken 65 min before surgery (baseline) and thereafter blood samples will be obtained 0 min., 15 min., 30 min., 45 min., 60 min., 90 min., 120 min., 180 min., 240 min., 300 min., 360 min. and 420 min. after administration of melatonin. Blood samples will be obtained again after administration of melatonin at 9 pm. in the evening in the same manner as described above. Plasma samples will be stored at minus 80 C and analyzed at the research laboratory of the Department of surgery, Herlev Hospital. The analysis will be preformed with the RIA-technique.

The second part is a randomized, double-blind, placebo-controlled study with a total of 32 participants divided into a intervention group (16) and a placebo group (16). In this part the investigators intend to investigate the anxiolytic and sleep-promoting effects of melatonin. Melatonin and placebo will be administrated at 9 pm. the evening before surgery, 120 min. before surgery, immediately after surgery in the PACU and at 9 pm the evening after surgery.

Anxiety will be measured by the State-Trait Anxiety Inventory (STAI) and a VAS-scale (0 mm = no anxiety and 100 mm = worst anxiety). Quality of sleep will be measured at the VAS-scale as well (0 mm = best sleep and 100 = worst sleep).

Randomization will be performed by a computer at randomization.com. The "first generator" function is used. The randomization will be preformed in blocks of 4 patients in each.

Manufacturing of medications and randomization will be made by an independent pharmacist.

The primary outcome is preoperative anxiety as measured on the STAI. A previous study investigated preoperative anxiety before hernia surgery and found a mean of 35.4 (SD 10.0) on the STAI scale. There does not exist any generally accepted measure of how large a change on the STAI scale constitutes a clinically important difference. However, a change equal to one standard deviation has been suggested. In the present study, this corresponds to a minimal relevant difference (MIREDIF) of 10 points on the STAI scale or 28%. A power of 80% was defined, a significance level of 5% and a minimal relevant difference (MIREDIF) of 28%. From these assumptions, 16 patients in each treatment group is needed

Statistics Anxiety and sleep quality will be compared at individual timepoints between groups Comparison will be performed either by Mann-whitheys-test or unpaired t-test, depending on the distribution of data. Values are considered significant at a p-value at 5% or less. Data will be reported as mean (SD) or median (IQR) depending on the distribution of data.

Data for the blood samples will be presented as AUC plasma concentrations, half-life, maximum concentration and time to maximum concentration.

ELIGIBILITY:
Inclusion Criteria part one:

* Patients who are candidates for breast surgery.
* BMI between 18 and 30
* Visible veins in the elbow region
* Fertile women use anti-contraception and have performed a negative pregnancy test

Exclusion Criteria part one:

* Patients, who use daily opioids, benzodiazepines or melatonin
* Patients diagnosed with a psychiatric disorder (defined as in medical treatment)
* Patients with severe physical disease (ASA 3-4)
* Patients with previous or ongoing alcohol or drug abuse
* Patients with liver disease (defined as in medical treatment)
* Patients diagnosed sleep disturbances
* Patients who are unable to cooperate according to the protocol
* Patients with allergy to melatonin

Inclusion Criteria part two:

- Male patients who are candidates for inguinal or umbilical hernia reapir

Exclusion Criteria part two:

* Patients, who use daily opioids, benzodiazepines or melatonin
* Patients diagnosed with a psychiatric disorder (defined as in medical treatment)
* Patients with severe physical disease (ASA 3-4)
* Patients with previous or ongoing alcohol or drug abuse
* Patients with liver disease (defined as in medical treatment)
* Patients diagnosed sleep disturbances
* Patients who are unable to cooperate according to the protocol
* Patients with allergy to melatonin

Withdrawal- and drop-out criteria part 2:

* Patients can withdraw at any time during trial
* Complications during surgery occur that lead to:

  1. Immediate reoperation
  2. Hospitalization to intensive care unit
* If it is considered in the best interest of the patients physical- and psychological health to withdraw from the trial

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-08; Primary Completion 2021-03 (Actual); Study Completion 2021-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis B Zetner, MD., Principal Investigator — Herlev Hospital, Herlev Ringvej 75, Herlev, Denmark
Locations (1):
- Herlev Hospital, Herlev, Denmark

REFERENCES:
- [Derived] Madsen BK, Zetner D, Moller AM, Rosenberg J. Melatonin for preoperative and postoperative anxiety in adults. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD009861. doi: 10.1002/14651858.CD009861.pub3. PMID 33319916

RESULTS

PARTICIPANT FLOW:
Groups:
- Melatonin: Melatonin 10 mg, gelatin capsules. Pharmacokinetic study: 10 mg x 2. In the morning before surgery and in the evening after surgery.
  Anxiolytic and analgesic study: 10 mg x 4. Evening the day before surgery, the morning before surgery, immediately after surgery and the evening after surgery.
  Melatonin: Gelatin capsules
Period: Overall Study
Arm/Group | Melatonin | Placebo
Started | 18 | 18
Completed | 16 | 17
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Melatonin | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 25
  >=65 years | 5 | 6 | 11
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [45 to 62] | 60 [50 to 69] | 59 [48 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 18 | 18 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 18 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 18 | 18 | 36
Hernia (inguinal/umbilical) [Count of Participants; unit: Participants]
  Inguinal hernia | 17 | 14 | 31
  Umbilical hernia | 1 | 4 | 5
Surgery (laparoscopic/open) [Count of Participants; unit: Participants]
  Laparoscopic | 17 | 13 | 30
  Open | 1 | 5 | 6
Baseline State anxiety (at enrolment) [Median (Inter-Quartile Range); unit: units on a scale] — The "State" scale of the State-Trait Anxiety Inventory (STAI). Construct: Current level of anxiety. Scale range: 20-40 (higher scores indicate higher level of current anxiety) Scores are calculated according to the STAI scoring manual by adding point from each item (possible point for each item is 1-4).
  units on a scale | 27 [22 to 34] | 27 [23 to 31] | 27 [22 to 33]
Baseline Trait anxiety (at enrolment) [Median (Inter-Quartile Range); unit: units on a scale] — The "Trait" scale of the State-Trait Anxiety Inventory (STAI). Construct: Inherent level of anxiety. Scale range: 20-40 (higher scores indicate higher level of inherent anxiety) Scores are calculated according to the STAI scoring manual by adding point from each item (possible point for each item is 1-4).
  units on a scale | 30 [23 to 34] | 27 [24 to 30] | 29 [23 to 32]
Baseline VAS anxiety [Median (Inter-Quartile Range); unit: units on a scale] — Visual analogue scale of anxiety. Construct: Current level of anxiety. Scale range: 1-10 (higher scores indicate higher level of current anxiety)
  units on a scale | 5 [0 to 10] | 5 [1 to 14] | 5 [1 to 13]

OUTCOME MEASURES:

1. Primary Outcome: Preoperative Anxiety
Description: The "State" scale of the State-Trait Anxiety Inventory (STAI). Construct: Current level of anxiety. Scale range: 20-40 (higher scores indicate higher level of current anxiety) Scores are calculated according to the STAI scoring manual by adding point from each item (possible point for each item is 1-4).
Time Frame: 60 minutes preoperative
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 16 | 17
score on a scale | 27 [24 to 34] | 28 [24 to 33]

2. Secondary Outcome: Postoperative Anxiety
Description: State-Trait Anxiety Index
Time Frame: at the preoperative interview, 60 minutes prior to surgery and 4 hours postoperatively.
Reporting Status: Not Posted

3. Secondary Outcome: Pre- and Postoperative Anxiety
Description: Visual analog scale
Time Frame: at the preoperative interview, 60 minutes prior to surgery, 1 and 4 hours postoperatively.
Reporting Status: Not Posted

4. Secondary Outcome: Intraoperative Requirement of Remifentanil
Description: µg/kg/min
Time Frame: intraopeative
Reporting Status: Not Posted

5. Secondary Outcome: Intraoperative Requirement of Propofol
Description: mg/kg/min
Time Frame: intraoperative
Reporting Status: Not Posted

6. Secondary Outcome: Use of Rescue-opioids in the PACU
Description: dose
Time Frame: 0-24 hours postoperative
Reporting Status: Not Posted

7. Secondary Outcome: Use of Rescue-opioids in the Ward
Description: dose
Time Frame: 0-24 hours postoperative
Reporting Status: Not Posted

8. Secondary Outcome: Perioperative Sleep Quality
Description: Visual analog scale
Time Frame: 24 hours
Reporting Status: Not Posted

9. Secondary Outcome: General Well-being and Fatigue
Description: Visual analog scale
Time Frame: 24 hours
Reporting Status: Not Posted

10. Secondary Outcome: Plasma Concentrations of Melatonin
Description: pg/ml
Time Frame: baseline, 0 min, 15 min, 30 min, 45 min, 60 min, 90 min, 120 min, 180 min, 240 min, 300 min, 360 min and 420 min. after melatonin administration.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | Melatonin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT02386319/Prot_SAP_000.pdf